CLINICAL TRIAL: NCT06160206
Title: A Phase II Open Label, Randomized Study Testing the Efficacy of Retifanlimab in Combination with Bevacizumab and Hypofractionated Radiotherapy in Patients with Recurrent GBM
Brief Title: Retifanlimab with Bevacizumab and Hypofractionated Radiotherapy for the Treatment of Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACCRU-NO-2301; NCI-2023-09550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-NO-2301 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Glioblastoma; Recurrent WHO Grade 4 Glioma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Retifanlimab, bevacizumab and HFRT) (Experimental): ARM I: Patients receive retifanlimab IV over 30 minutes on day 1 and bevacizumab IV on day 1 and 15 of each cycle. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo HFRT QD, starting in cycle 1 on day 15 for 10 treatments. Patients undergo MRI or CT, as well as blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Biological: Retifanlimab
- Arm B (Bevacizumab and radiation) (Experimental): Patients receive bevacizumab IV on day 1 and 15 of each cycle. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo HFRT QD, starting in cycle 1 on day 15 for 10 treatments. Patients undergo MRI or CT, as well as blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; CT-P16; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Ancillary studies
Radiation: Hypofractionated Radiation Therapy — Undergo radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Biological: Retifanlimab — Given IV
  Other Names: INCMGA 0012; INCMGA-0012; INCMGA00012; INCMGA0012; MGA 012; MGA-012; MGA012; Retifanlimab-dlwr; Zynyz
  Arms: Arm A (Retifanlimab, bevacizumab and HFRT)

SUMMARY:
This phase II trial tests how well retifanlimab with bevacizumab and hypofractionated radiotherapy, compared to bevacizumab and hypofractionated radiotherapy alone, works in treating patients with glioblastoma that has come back after a period of improvement (recurrent). A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as retifanlimab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Giving retifanlimab with bevacizumab and hypofractionated radiotherapy may work better in treating patients with recurrent glioblastoma than bevacizumab and hypofractionated radiotherapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the overall survival at 9 months (OS-9) of the combination of retifanlimab, bevacizumab and hypofractionated radiation therapy (HFRT) vs. the control group treated with bevacizumab and HFRT.

SECONDARY OBJECTIVES:

I. To assess the overall survival (OS) in this patient population for each regimen.

II. To assess the progression free survival (PFS) in this patient population for each regimen.

III. To assess the objective response rate (ORR) in this patient population for each regimen.

IV. To assess the neurologic function by Neurologic Assessment in Neuro-Oncology (NANO) in this patient population for each regimen.

V. To assess the frequency and severity of adverse events in this patient population for each regimen.

CORRELATIVE OBJECTIVE:

I. To assess the anti-glioma immune response before and after retifanlimab including assessment of immune cells phenotyping, function and activation in the pre-/post-treatment blood, and changes in cytokine levels over time.

OUTLINE: Patients are randomized to 1 of 2 arms

ARM A: Patients receive retifanlimab intravenously (IV) over 30 minutes on day 1 and bevacizumab IV on day 1 and 15 of each cycle. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo HFRT once daily (QD), starting in cycle 1 on day 15 for 10 treatments. Patients undergo magnetic resonance imaging (MRI) or computed tomography (CT), as well as blood sample collection throughout the study.

ARM B: Patients receive bevacizumab IV on day 1 and 15 of each cycle. Treatment repeats every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo HFRT QD, starting in cycle 1 on day 15 for 10 treatments. Patients undergo MRI or CT, as well as blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days. Survival follow-up is every 2 months for the first year, and then every 6 months for up to 4 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Recurrent World Health Organization (WHO) grade IV glioblastoma. Note: Any number of recurrences are allowable. Glioblastoma (GBM) variants and molecular GBM are allowed
* Candidates for radiotherapy
* Prior use of bevacizumab is allowed as long as the last treatment is > 4 months prior to randomization
* Dexamethasone dose ≤ 4mg daily at the time of randomization (higher dose of steroid for symptom control is allowed during the study)
* Karnofsky performance status ≥ 60%
* Measurable disease or non-measurable disease per Response Assessment in Neuro-Oncology (RANO) criteria
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3 (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the Academic and Community Cancer Research Untied (ACCRU) website under "General Forms"
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Creatinine ≤ 1.5 x ULN (obtained ≤ 28 days prior to registration)

  * NOTE: If your site laboratory reports use different units of measurement than what is required by the protocol eligibility requirements, please use the "Lab Test Unit Conversion Worksheet" available on the ACCRU website under "General Forms"
* Negative pregnancy test done ≤ 14 days prior to registration for women of childbearing potential only. (Pregnancy test can be urine or serum.)

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
  * A female of childbearing potential is a sexually mature female who:

    * 1) Has not undergone a hysterectomy or bilateral hysterectomy; or
    * 2) Has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months)
* Provide informed written consent ≤ 28 days prior to registration
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study, i.e., active treatment)
* Willing to provide mandatory blood specimens for correlative research purposes

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception (men and women)
* Co-morbid systemic illness or other severe concurrent disease which, in the judgement of the investigator, would make the patient inappropriate for entry into the study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Receiving any other investigational agent which would be considered treatment for the primary neoplasm ≤ 2 weeks prior to registration
* Active uncontrolled autoimmune disease or syndrome (i.e. moderate or severe rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, active inflammatory bowel disease) that has required systemic treatment in the past 2 years (i.e. with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs) or who are receiving systemic therapy for an autoimmune or inflammatory disease (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Subjects are permitted to enroll if they have vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Has a severe acute or chronic medical condition including immune colitis, inflammatory bowel disease (may be enrolled at the discretion of the principal investigator [PI]), immune pneumonitis, or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to epacadostat, retifanlimab, bevacizumab, or other agents used in the study
* Has had an allogeneic tissue/solid organ transplant
* Has uncontrolled human immunodeficiency virus (HIV) (HIV ½ antibodies). Well-controlled HIV is defined as CD4+ count > 300 cells, undetectable viral load, and receiving highly active antiretroviral therapy (HAART)/antiretroviral therapy (ART). Study specific HIV testing is not required for patients who do not have any prior history of HIV
* Has uncontrolled active hepatitis B (HBV) (e.g., hepatitis B serum antigen [HBsAg] reactive or HBV dioxyribonucleic acid [DNA] detected by quant real time polymerase chain reaction [RT PCR]) or hepatitis C (e.g. hepatitis C serum antigen [HCsAg] reactive or hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative or quantitative] is detected)
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Time until death from any cause, assessed up to 9 months after registration
  Defined as the proportion of patients who are alive 9 months after randomization based on Kaplan Meier estimate. The proportion of patients alive will be compared between treatment arms using a z-score test statistic. The 9-month OS Kaplan Meier estimate and corresponding 95% confidence interval for each arm will be reported.

SECONDARY OUTCOMES:
OS | Up to 4 years after registration
  Overall survival is defined as the time from registration to death from any cause. OS will be estimated using the Kaplan-Meier method. The logrank test will be used to compare the distribution between treatment arms. The median OS and corresponding 95% confidence interval (by Brookmeyer and Crowley) will be reported for each treatment arm.
Progression free survival (PFS) | Up to 4 years after registration
  Progression free survival is defined as the time from randomization to documentation of disease progression or death due to any cause, whichever is first. The distribution of PFS will be estimated using the method of Kaplan-Meier. PFS will be compared between the 2 treatment arms using the log-rank test. The median PFS and corresponding 95% confidence intervals will be reported.
Objective response rate (ORR) | Up to 4 years after registration
  Objective response is defined as experiencing a complete response (CR) or partial response (PR) (as defined by RANO criteria, see section 11.0) while on protocol treatment. Objective response rate (ORR) is defined as the number of patients who experience objective response divided by the number of patients in the primary analysis population. ORR will be compared between the 2 treatment arms. Confidence intervals for ORR will be calculated according to the approach of Clopper and Pearson. Overall response rate and the corresponding 95% confidence interval will be reported.
Neurologic function domain scores | Up to 2 months after registration
  Neurologic function domain scores of the Neurologic Assessment in Neuro-Oncology be summarized by descriptive statistics including mean, median, standard deviation, and range for each regimen at each time point. The difference between baseline and 2 months (1st restaging scan) will be compared using a Wilcoxon Rank Sum test across arm for each domain. The median difference for each domain and 1st and 3rd quartile will be reported for each arm.
Incidence of adverse events | Up to 4 years after registration
  The overall adverse event rates for grade 3 or higher adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jian L Campian, Principal Investigator — Academic and Community Cancer Research United
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota